CLINICAL TRIAL: NCT05747066
Title: Nutritional Intake, Nutritional Status and Physical Activity Level in People Who Have Undergone a Major Dysvascular Lower Limb Amputation
Brief Title: Nutrition in People With a Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 10929
Record Dates: First submitted 2023-01-23; First posted 2023-02-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Diet, Food, and Nutrition; Nutrition Disorders; Amputation
Keywords: Nutrition; Malnutrition; Physical activity; Amputation; Outcomes
MeSH Terms: conditions — Nutrition Disorders; Malnutrition; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this prospective longitudinal observational cohort study is to determine the nutritional intake, nutritional status, and physical activity level in people who have undergone a major dysvascular lower limb amputation (LLA) at different moments post-LLA (during hospital admission several days post-LLA, and at 5 weeks, 6 months, and 9 months post-LLA). The main questions this study aims to answer are:

* What is the nutritional intake, nutritional status, and physical activity level at different moments post-LLA?
* What is the association between nutritional intake and physical activity level, and nutritional status?
* What is the association between nutritional intake, nutritional status and physical activity level and clinical outcomes (mortality, wound healing, quality of life, physical functioning)?

DETAILED DESCRIPTION:
People requiring an LLA are at high risk for adverse clinical outcomes. Undernutrition and low physical activity level may affect clinical outcomes negatively. However, little is known about the nutritional intake, nutritional status and physical activity level in the LLA population, and their association with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing or recently (i.e., within the last seven weeks) having undergone a major dysvascular lower limb amputation (i.e., Syme amputation or more proximal level)
* 18 years or older
* Able to collaborate

Exclusion Criteria:

* Requiring re-amputation
* Severe malabsorption disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of people who have undergone a major dysvascular lower limb amputation.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Nutritional intake at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Nutritional intake will be assessed by a 24h recall. Nutritional intake includes intake of energy, protein, carbohydrates, and fat, and will be classified as adequate/inadequate intake.
Diet quality at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  The Dutch Healthy Diet Index will be calculated on the data of the 24h recall. The 15 components of the Dutch Healthy Diet Index represent the 15 food-based Dutch dietary guidelines of 2015. The score ranges from 0 to 10 for each component, giving a total score between 0 (no adherence) and 150 (complete adherence).
Patient-Generated Subjective Global Assessment at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Nutritional status will be determined based on the use of the Patient-Generated Subjective Global Assessment (PG-SGA). Completing the PG-SGA will result in a numerical score (0-52), as well as categorization of nutritional status (PG-SGA Stage A = well nourished, PG SGA Stage B = moderate or suspected undernutrition, PG-SGA Stage C = severely undernourished).
Muscle mass at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Muscle mass will be determined by measuring the mid-upper arm circumference and the triceps skinfold, in mm.
Muscle strength at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Muscle strength will be determined by the handgrip strength, in kgf.
Body mass index at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Body mass index will be determined based on weight and height, and adjusted for LLA level, in kg/m^2.
Physical activity level by Activ8 accelerometer at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Physical activity level will be determined based on data from the Activ8 accelerometer. The Activ8 is a tri-axis accelerometer (2M Engineering, Valkenswaard, The Netherlands) which determines the time spent lying/sitting, standing, walking, running, and cycling for at least 3 consecutive days. The following outcome variables will be calculated: percentage of time spent active, intensity of behavior (counts/min), average number of active bouts, and mean duration of active bouts.
Physical activity level by adapted Short QUestionnaire to ASsess Health-enhancing physical activity at each time point and change over time | During hospital admission 2 to 12 days post-LLA, at 5 weeks post-LLA, at 6 months post-LLA, at 9 months post-LLA
  Physical activity level will be determined based on the adapted Short QUestionnaire to ASsess Health-enhancing physical activity (Adapted-SQUASH). The Adapted-SQUASH is a 19-item self-reported recall questionnaire designed to assess physical activity among persons with disabilities. Total activity score will be calculated (minutes x intensity) together with total minutes of activity/week, and total minutes of light, moderate or vigorous activity/week.

SECONDARY OUTCOMES:
Mortality | Through study completion, up to 9 months post-LLA
  Data regarding mortality will be collected from the Statistics Netherlands (Dutch: Centraal Bureau voor de Statistiek).
Wound healing | At 5 weeks post-LLA
  Wound healing will be classified as healed wound or open wound. Healed wound is defined as closed wound, i.e., skin is intact and the underneath tissue is not exposed. Furthermore, the TIME criteria will be assessed.
Quality of life assessed by World Health Organization Quality of Life Questionnaire - BREF at each time point and change over time | At 5 weeks, and 6 and 9 months post-LLA
  Quality of life will be assessed by the World Health Organization Quality of Life Questionnaire - BREF. This is a self-reported instrument. Possible scores range from 0 to 100. A higher score indicates a better quality of life.
K-level at each time point and change over time | At 6 and 9 months post-LLA
  Potential level of functioning will be assessed using the K-level.
6-minute walk test at each time point and change over time | At 6 and 9 months post-LLA
  Physical functioning will be assessed by the 6-minute walk test. More distance covered during the 6-minute walk test indicates a better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Jan HB Geertzen, Principal Investigator — University Medical Center Groningen
Locations (6):
- Netherlands (6):
  - Treant Zorggroep, Emmen, Drenthe
  - Isala Zwolle, Zwolle, Overijssel
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Martini Ziekenhuis Groningen, Groningen, Provincie Groningen
  - Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen
  - Ommelander Ziekenhuis Groep, Scheemda, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided